CLINICAL TRIAL: NCT05690451
Title: The Role of Non-contrast Abbreviated MRI for Secondary Surveillance of Hepatocellular Carcinoma After Curative Treatment: a Prospective Multicenter Study
Brief Title: Non-contrast Abbreviated MRI for Secondary Surveillance of HCC
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Lee, Clinical professor, Seoul National University Hospital
Other Study IDs: H-2106-183-1230; KCT0006395 (Registry Identifier: https://cris.nih.go.kr/)
Record Dates: First submitted 2022-12-28; First posted 2023-01-19 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Secondary surveillance of hepatocellular carcinoma; Contrast enhanced liver CT; non-contrast abbreviated MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: non-contrast abbreviated MRI — Liver MRI without contrast injection. The following sequences will be obtained from all of the participants.
  * Axial heavily and regular T2 WI
  * precontrast fat-suppressed T1 WI
  * Diffusion-weighted image using b-value of 0, 50 or 400, and 800 or 1000
Diagnostic Test: Contrast enhanced liver CT — Liver CT with iodine contrast injection This test will be served as a standard diagnostic test. The following phases will be obtained
  * precontast, arterial phase, portal venous phase and delayed phase

SUMMARY:
This prospective multicenter study aimed to compare the diagnostic performance of non-contrast abbreviated MRI in detecting recurrent HCC after curative treatment to that of contrast-enhanced liver CT.

DETAILED DESCRIPTION:
This study was designed as a prospective single-arm intra-individual comparison multicenter study

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-year old and 85-year old
* Patients with a history of curative treatment for HCC including surgical resection or local ablation
* No recurrence after curative treatment of HCC for more than two years
* Patient who has the plan to perform contrast-enhanced liver CT for secondary surveillance for HCC (i.e., to detect de novo or recurrent HCC)

Exclusion Criteria:

* Estimated GFR less than 60
* Previous history of severe allergic reaction to the iodinated contrast agent
* Patients with claustrophobia who can't undergo MR examination
* Patients having cochlear implants or cardiac pacemaker

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent curative treatment for HCC including surgical resection or local ablation and have a more than a two-year disease-free period, needing continuous surveillance for the development of HCC will be candidates for this study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Accuracy per patient | Within 6 months from the study completion
  Accuracy for detection of recurrent HCC per patient

SECONDARY OUTCOMES:
Specificity per patient | Within 6 months from the study completion
  Specificity for detection of recurrent HCC per patient
Sensitivity per patient | Within 6 months from the study completion
  Sensitivity for detection of recurrent HCC per patient

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ho Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam, Korea (the Republic Of)
  - Asan Medical Center, Seoul, Korea (the Republic Of)
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) of this study will be available for reasonable requests after approval of IRB